CLINICAL TRIAL: NCT00893542
Title: A Single Dose, 2-Period, 2-Treatment 2-Way Crossover Bioequivalency Study of Mycophenolate Mofetil 250 mg Capsules Under Fasting Conditions
Brief Title: Bioequivalency Study of Mycophenolate Mofetil 250 mg Capsules Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MYCO-C250-PVFS-1
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Prophylaxis of Organ Rejection
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mycophenolate Mofetil — mycophenolate mofetil 250 mg capsule
  Other Names: CellCept

SUMMARY:
The objective of this study was to prove the bioequivalence of Mycophenolate Mofetil 250 mg Capsules under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C. Treatment with known enzyme altering drugs. History of allergic or adverse response to mycophenolate mofetil or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2005-11; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | baseline, 2-period, 14 day washout

CONTACTS AND LOCATIONS:
Overall Officials: William Allen Alexander, M.D., Principal Investigator — CEDRA Clinical Research, LLC
Locations (1):
- CEDRA Clinical Research, LLC, Austin, Texas, United States